CLINICAL TRIAL: NCT03035175
Title: A Randomized Control Trial: Does Guidance Using Video Laryngoscopy Improve Residents' Success in Neonatal Intubation?
Brief Title: Using Video Laryngoscopy for Neonatal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RSRB00051876
Record Dates: First submitted 2017-01-24; First posted 2017-01-27 (Estimated); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Education, Medical
Keywords: Residences; Video Laryngoscopy; Intubations; Neonatal; NICU; neonates; Medical Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Laryngoscopy Group (Experimental): Subjects enrolled in this arm received real-time guidance from a supervisor utilizing the screen of the video laryngoscope while the subjects performed direct neonatal intubations in the NICU.
  Interventions: Other: Video Laryngoscopy
- Traditional Laryngoscopy Group (Active Comparator): Subjects enrolled in this arm, received traditional guidance while they performed direct neonatal intubations in the NICU.
  Interventions: Other: Traditional Laryngoscopy

INTERVENTIONS:
Other: Video Laryngoscopy — Residents intubate using video laryngoscopy.
  Other Names: Technology-Assisted Instruction
  Arms: Video Laryngoscopy Group
Other: Traditional Laryngoscopy — Residents intubate without using video laryngoscopy.
  Other Names: Traditional Instruction
  Arms: Traditional Laryngoscopy Group

SUMMARY:
This study examines the effectiveness of utilizing video laryngoscopy to give real-time guidance during neonatal intubations to improve residents' success at performing intubations.

DETAILED DESCRIPTION:
To evaluate whether residents who receive guidance from a supervisor concurrently viewing the neonate's airway via video laryngoscopy will have a higher rate of successful neonatal intubations than residents receiving guidance using traditional direct laryngoscopy.

The investigators conducted a randomized controlled trial involving 48 first and second year pediatric and medicine-pediatric residents who received either video-facilitated (VDL) or traditional (TDL) supervisor guidance during direct laryngoscopy. Residents attempted intubations in the neonatal intensive care unit according to their randomization group. The primary outcome was a successful intubation that occurred within two attempts.

ELIGIBILITY:
Inclusion Criteria:

* 1st and 2nd Year Pediatric and Medicine-Pediatric Residents at the University of Rochester

Exclusion Criteria:

* Residents who declined participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-05; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of Successful Intubations | 12 months
  A successful intubation is defined as the placement of an endotracheal tube in the infant's trachea within two attempts.

SECONDARY OUTCOMES:
Number of successful intubations by resident year | 12 months
Number of residents with successful intubations on the first and subsequent patients | 12 months
Average length of time of intubation attempts | 12 months
Number of both serious and non-serious adverse events | 12 months
Number of successful intubations by residency program | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rita Dadiz, DO, Principal Investigator — University of Rochester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haubner LY, Barry JS, Johnston LC, Soghier L, Tatum PM, Kessler D, Downes K, Auerbach M. Neonatal intubation performance: room for improvement in tertiary neonatal intensive care units. Resuscitation. 2013 Oct;84(10):1359-64. doi: 10.1016/j.resuscitation.2013.03.014. Epub 2013 Apr 3. PMID 23562374
- [Background] Falck AJ, Escobedo MB, Baillargeon JG, Villard LG, Gunkel JH. Proficiency of pediatric residents in performing neonatal endotracheal intubation. Pediatrics. 2003 Dec;112(6 Pt 1):1242-7. doi: 10.1542/peds.112.6.1242. PMID 14654592
- [Background] O'Shea JE, Thio M, Kamlin CO, McGrory L, Wong C, John J, Roberts C, Kuschel C, Davis PG. Videolaryngoscopy to Teach Neonatal Intubation: A Randomized Trial. Pediatrics. 2015 Nov;136(5):912-9. doi: 10.1542/peds.2015-1028. Epub 2015 Oct 19. PMID 26482669
- [Background] Moussa A, Luangxay Y, Tremblay S, Lavoie J, Aube G, Savoie E, Lachance C. Videolaryngoscope for Teaching Neonatal Endotracheal Intubation: A Randomized Controlled Trial. Pediatrics. 2016 Mar;137(3):e20152156. doi: 10.1542/peds.2015-2156. Epub 2016 Feb 12. PMID 26908701